CLINICAL TRIAL: NCT03201744
Title: Prospective Randomized Trial of Moderate vs Deep Neuromuscular Blockade During Laparoscopic Ventral Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Konstantinos Spaniolas, Associate Professor of Surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1034023-3
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hernia, Ventral; Neuromuscular Blockade; Pneumoperitoneum
MeSH Terms: conditions — Hernia, Ventral; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Neuromuscular Block (Experimental): Train of four count of 1-2. All procedures will start with low-pressure insufflation (8 mm Hg). Surgeon assessment of the conditions will be serially performed during surgery on an established visual scale. If conditions are deemed less than adequate (score 1-2), insufflation pressure will incrementally increase up to 15 mm Hg. Reversal of muscle relaxation will be performed at the end of the procedure using established medications used in clinical practice. In theory, deep relaxation may require a more prolonged reversal process, but using contemporary medical agents (sugammadex), reversal from deep relaxation is prompt (2-3 minutes) without any additional delays.
  Interventions: Procedure: Patients will be randomized to moderate (TOF 1-2) or deep (post tetanic count 1-2) relaxation. Low pressure insufflation (start pressure set at 8 mm Hg)
- Deep Neuromuscular Block (Experimental): Post tetanic count of 1-2. All procedures will start with low-pressure insufflation (8 mm Hg). Surgeon assessment of the conditions will be serially performed during surgery on an established visual scale. If conditions are deemed less than adequate (score 1-2), insufflation pressure will incrementally increase up to 15 mm Hg. Reversal of muscle relaxation will be performed at the end of the procedure using established medications used in clinical practice. In theory, deep relaxation may require a more prolonged reversal process, but using contemporary medical agents (sugammadex), reversal from deep relaxation is prompt (2-3 minutes) without any additional delays.
  Interventions: Procedure: Patients will be randomized to moderate (TOF 1-2) or deep (post tetanic count 1-2) relaxation. Low pressure insufflation (start pressure set at 8 mm Hg)

INTERVENTIONS:
Procedure: Patients will be randomized to moderate (TOF 1-2) or deep (post tetanic count 1-2) relaxation. Low pressure insufflation (start pressure set at 8 mm Hg) — All procedures will start with low insufflation pressure (8 mmHg). Surgical field assessment (scale 1-5) will be performed every 5 minutes (Martini Br J Anaesth 2014). If conditions are poor (rating 1-2), intraperitoneal insufflation will be incrementally increased (10 mmHg, 12 mmHg, 15 mmHg) every 5 minutes as needed.Reversal of muscle relaxation will be performed at the end of the procedure using established medications used in clinical practice. In theory, deep relaxation may require a more prolonged reversal process, but using contemporary medical agents (sugammadex), reversal from deep relaxation is prompt (2-3 minutes) without any additional delays.

SUMMARY:
The proposed study aims to assess the effect of different levels of muscle relaxation on the success of low-pressure insufflation, surgical conditions and patient recovery following laparoscopic repair of a ventral hernia (VHR) between 2 and 10cm in diameter. Patients will be randomized to moderate (TOF 1-2) or deep (post tetanic count 1-2) relaxation.

Specific Aim 1. Compare two different modes of neuromuscular blockade (moderate and deep) on the ability to maintain low insufflation pressure during laparoscopic VHR. All procedures will start with low-pressure insufflation (8 mm Hg). Surgeon assessment of the conditions will be serially performed during surgery on an established visual scale. If conditions are deemed less than adequate (score 1-2), insufflation pressure will incrementally increase up to 15 mm Hg. Outcome for this specific aim will be the mean insufflation pressure during each procedure, and the ability to perform low-pressure laparoscopic VHR.

Specific Aim 2. Evaluate the success of moderate neuromuscular blockade on the ability to maintain good conditions (visual scale grade 4 or 5) for each. Surgical conditions will be considered successful when scores are maintained at 4 or 5 throughout the duration of the procedure. Outcome for this aim will be the mean score for surgical condition assessment for each procedure, using a previously published surgeon-driven scoring system (score 4-5 will be used as a surrogate of good visualization).

Specific Aim 3. Assess patient recovery with low and high insufflation pressures during laparoscopic VHR. Patient overall satisfaction with recovery, pain level, pain medication requirement, PONV incidence and severity will be assessed in multiple time points following surgery. Outcomes for this aim will be mean pain (visual scale), PONV severity (analogue score) and incidence (binary outcome), and patient satisfaction using the QoR-15 survey. Assessments will be performed at 30 minutes, 1, 12 and 24 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-75 years old
* Umbilical, ventral, epigastric, spigelian or incisional hernia
* Plan for laparoscopic ventral hernia repair with mesh
* Estimated fascial defect between 2-10 cm in maximum diameter

Exclusion Criteria:

* Allergy to medications delineated in the protocol (muscle blockade, anesthetics, reversal agents)
* Inability to provide informed consent
* Body mass index of 35 or over
* Multiple recurrent hernias (>1)
* Creatinine clearance < 30 ml/min (using the Cockcroft-Gault calculation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Mean insufflation pressure during each procedure as a continuous variable | will be assessed every 5 minutes during surgery (while subject is undergoing laparoscopic ventral hernia repair)

SECONDARY OUTCOMES:
Surgical condition assessment | every 5 minutes during surgery (while subject is undergoing laparoscopic ventral hernia repair)
PONV severity (analogue score) and incidence (binary) | it will be assessed at 30 minutes, 1 hour, 12 hours and 24 hours after the completion of laparoscopic ventral hernia repair
Patient satisfaction (QoR-15). | it will be assessed 24 hours after the completion of laparoscopic ventral hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Spaniolas, MD, Principal Investigator — StonyBrook University Hospital
Locations (1):
- Shabana Humayon, Stony Brook, New York, United States